CLINICAL TRIAL: NCT03500848
Title: Sirolimus-based Immunosuppression Treatment Regimen for Liver Transplantation: A Multicenter, Open-label, Randomized, Controlled Clinical Trial in Liver Transplant Recipients With Hepatocellular Carcinoma
Brief Title: Sirolimus-based Immunosuppression Treatment Regimen for Liver Transplantation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southern Medical University, China (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Chongyang Duan, Post-doctoral Fellow, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-GDEK-001
Record Dates: First submitted 2018-03-29; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; Sirolimus; Tacrolimus; HCC recurrence free survival
MeSH Terms: interventions — Tacrolimus; Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus-based group (Active Comparator): Tacrolimus-based immunosuppression regimen: Tacrolimus+MMF and/or steroids
  Interventions: Drug: Tacrolimus; Drug: MMF and/or steroids
- Sirolimus-based group (Experimental): Sirolimus-based immunosuppression regimen: Tacrolimus (Tacrolimus elimination 30 (± 5) days post LT)+Sirolimus+MMF and/or steroids
  Interventions: Drug: Tacrolimus (Tacrolimus elimination); Drug: Sirolimus; Drug: MMF and/or steroids

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus will be started between 3 and 7 days post-transplantation and continued after randomization at a dose of 1.0 mg twice a day (bid, 2 mg daily dose). The tacrolimus trough level is measured twice a week for 1 month, followed by trough level once a month thereafter. Tacrolimus trough levels are targeted to be maintained at 8-15ng/ml until Month 6. After Month 6, the dose will be adjusted over time to maintain steady-state tacrolimus trough blood levels of approximately 5-10 ng/mL.
  Other Names: FK-506; Fujimycin; Prograf; Protopic; Advagraf
  Arms: Tacrolimus-based group
Drug: Tacrolimus (Tacrolimus elimination) — Tacrolimus will be started between 3 and 7 days post-transplantation at a dose of 1.0 mg twice a day (bid, 2 mg daily dose) for 30 (± 5) days and eliminated when randomization is done.
  Other Names: FK-506; Fujimycin; Prograf; Protopic; Advagraf
  Arms: Sirolimus-based group
Drug: Sirolimus — Within 24 hours of randomization, sirolimus will be started at a dose of 2.0 mg once a day. The sirolimus trough level is measured twice a week for 1 month, followed by trough level once a month thereafter. The dose will be adjusted over time to maintain steady-state sirolimus trough blood levels of approximately 4-10 ng/mL.
  Other Names: Rapamune
  Arms: Sirolimus-based group
Drug: MMF and/or steroids — For patients in both groups, MMF and/or steroids are initiated at or prior to the time of liver transplantation according to local practice. Steroids reduction is encouraged by 3 months post liver transplantation.
  Other Names: Mycophenolate mofetil

SUMMARY:
This is a multicenter, open-label, randomized, controlled clinical trial, in order to compare sirolimus-based (tacrolimus-free) versus tacrolimus-based (sirolimus-free) immunosuppression regimen for Hepatocellular Carcinoma (HCC) patients after liver transplantation.

DETAILED DESCRIPTION:
This 5-year study consisted of a 2-year enrolment period and a 3-year follow-up period. Patients will be screened for eligibility prior to liver transplantation. Patients who have undergone successful liver transplantation will be initiated on a tacrolimus-based regimen that includes MMF and/or Steroids and enter the baseline period (between 3 and 7 days post-transplantation). At 30 (± 5) days post-transplantation, patients who meet additional randomization inclusion/exclusion criteria will be randomized into 2 groups of this study. In the first group, patients will be maintained on a tacrolimus-based (sirolimus-free) immunosuppression regimen. The second group will be treated with sirolimus-based (tacrolimus-free) immunosuppression regimen. For patients in both groups, mycophenolic acid prodrugs like mycophenolate mofetil (MMF) and steroids are initiated at the time of liver transplantation according to local practice. Steroids reduction is encouraged by 3 months post liver transplantation.

In the first year after randomization all patients will be followed up after month 1, 2, 3, 4, 5, 6, 8, 10 and 12. After that, patients are followed every 3 months. Tacrolimus and sirolimus trough levels in patients of both groups will be tested and adjusted if need be at each follow-up date to achieve the desired steady-state trough levels.

The primary endpoint is defined as HCC recurrence-free time interval between the date of liver transplantation and the date of HCC recurrence or death; patients who are alive and recurrence-free at the end of month 36 will be censored at the time of their last follow-up date. HCC recurrence can be determined during the entire follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Recipients who are 18-65 years of age
* Histologically proven HCC before randomization
* Recipients who have been initiated on an immunosuppressive regimen that contains tacrolimus, 3-7 days post-transplantation
* Allograft is functioning at an acceptable level by the time of randomization as defined by protocol specific laboratory values
* Ability and willingness to provide written informed consent and adhere to study regimen

Exclusion Criteria:

* Patients with non-HCC malignancies within the past 5 years
* Patients who are multiple-organ recipients
* Patients who are known HIV-positive patients
* Patients who have received mTOR inhibitors prior to day 30 after liver transplantation
* Patients with a known hypersensitivity to the drugs used on study or their class, or to any of the excipients
* Patients who have any surgical or medical condition, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and excretion of study drug
* Patients with a psychologic, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
HCC recurrence free survival | Randomization to Month 36
  The primary endpoint is defined as HCC recurrence-free time interval between the date of liver transplantation and the date of HCC recurrence or death; patients who are alive and recurrence-free at the end of month 36 will be censored at the time of their last follow-up date. HCC recurrence can be determined during the entire follow-up period.

SECONDARY OUTCOMES:
Overall survival | Randomization to Month 36
  Overall survival was defined as the time from date of randomization to date of death from any cause. If a patient was not known to have died, patient overall survival was censored as the date of last contact.
Incidence of acute rejection | Randomization to Month 36
  Incidence of acute rejection will be assessed in both groups.
Treatment failures defined as introduction of Tacrolimus to experimental group | Randomization to Month 36
  Treatment failures defined as introduction of Tacrolimus to experimental group
Graft survival | Randomization to Month 36
  Graft survival was defined as the time from the date of randomization to the date of graft loss. If a patient was not known to suffer from a graft loss or died without graft loss, time to graft loss was censored with date of last contact or date of death, respectively.
Incidence of adverse events | Randomization to Month 36
  Evaluation of common post Liver Transplantation Adverse Events: wound healing, bone marrow depression, hyperlipidemia, proteinuria, diabetes mellitus, diagnosed hypertension, infections.

CONTACTS AND LOCATIONS:
Overall Officials: Kebo Zhong, M.D, Principal Investigator — Department of Heptobiliary Surgery II, Zhujiang Hospital, Southern Medical University, China
Locations (3):
- China (3):
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital, Sun Yat-Sen University, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided